CLINICAL TRIAL: NCT03220594
Title: Serum Antimullerian Hormone Levels in Patients Who Underwent Hypogastric Artery Ligation
Brief Title: Serum AMH Levels in Patients Who Underwent Hypogastric Artery Ligation
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, MD,ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 1826
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: AMH
Keywords: hypogastric artery; anti-mullerian hormone; ovarian reserve; postpartum
MeSH Terms: interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypogastric artery ligation (HAL): Patients who underwent only hypogastric artery ligation performed during the delivery of their babies. Six months after the operation they will evaluated for their ovarian reserve via hormones and astral follicle count (AFC)
  Interventions: Procedure: hypogastric artery ligation
- HAL and hysterectomy: Patients who underwent both hypogastric artery ligation and hysterectomy performed during the delivery of their babies. Six months after the operation they will evaluated for their ovarian reserve via hormones and astral follicle count (AFC)
  Interventions: Procedure: hypogastric artery ligation
- Postpartum: Postpartum control group constituted of patients delivered baby without any complication and evaluated 6 months later.

INTERVENTIONS:
Procedure: hypogastric artery ligation — hypogastric artery ligation is the ligation of the internal iliac artery to stop bleeding related to obstetrics obstetric hemorrhage Hysterectomy is the removal of the uterus if bleeding can't stop by hypogastric artery ligation
  Other Names: hysterectomy
  Groups: HAL and hysterectomy; Hypogastric artery ligation (HAL)

SUMMARY:
To observe the effects of hypogastric artery ligation on serum antimullerian hormone levels.

DETAILED DESCRIPTION:
To measure and compare serum antimullerian hormone levels in patients who underwent hypogastric artery ligation/ hypogastric artery ligation+ hysterectomy and postpartum control. The procedures performed as an emergency life saving method during delivery. The reasons for hypogastric artery ligation/ hypogastric artery ligation+ hysterectomy were obstetric hemorrhage mainly uterine atony.

The serum levels of antimullerian hormone were measured 6 months after the operations and compared with matching postpartum controls. Serum levels of FSH, LH, PRL and TSH were also measured 6 months after the operation. Further, antral follicle count measured along with the aforementioned blood tests.

ELIGIBILITY:
Inclusion Criteria:

* age 18- 40 years
* no systemic or endocrine diseases
* patients who had hypogastric artery ligation and/or hysterectomy
* healthy postpartum patients as controls

Exclusion Criteria:

* history of chemotherapy and/or radiotherapy
* Obese patients
* patients with previous/present endometriosis
* patients with PCOS

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants are females undergoing delivery of their baby
Study Population: Patients who had hypogastric artery ligation and/or hysterectomy during their delivery. Control group is age-matched postpartum patients.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve | 6 months
  To evaluate postoperative ovarian reserve using anti-mullerian hormones and other ovary related hormones including FSH,LH

CONTACTS AND LOCATIONS:
Overall Officials: Alev Atıs, MD,ObGyn, Study Director — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of total abdominal hysterectomy on serum anti-Müllerian hormone levels: a pilot study — https://www.ncbi.nlm.nih.gov/pubmed/22268398
- See also: Effect of internal iliac artery ligation on ovarian blood supply and ovarian reserve — https://www.ncbi.nlm.nih.gov/pubmed/20128664